CLINICAL TRIAL: NCT05261399
Title: A Phase III, Randomised, Open-Label Study of Savolitinib in Combination With Osimertinib Versus Platinum-Based Doublet Chemotherapy in Participants With EGFR Mutated, MET-Overexpressed and/or Amplified, Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Progressed on Treatment With Osimertinib (SAFFRON).
Brief Title: Savolitinib Plus Osimertinib Versus Platinum-based Doublet Chemotherapy in Participants With Non-Small Cell Lung Cancer Who Have Progressed on Osimertinib Treatment
Acronym: SAFFRON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5087C00001; 2024-511169-12-00 (Registry Identifier: CTIS); 2021-006374-24 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-03-02 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma; Non-Small-Cell Lung
Keywords: Savolitinib; Osimertinib; EGFR; Amplified; Metastatic; MET Driven; carcinoma; NSCLC; overexpressed
MeSH Terms: conditions — Carcinoma; Neoplasm Metastasis | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; osimertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): Pemetrexed (500 mg/m2) with either cisplatin (75 mg/m2) or carboplatin (AUC5) on Day 1 of 21-day cycles (Q3W) for 4 cycles, followed by pemetrexed maintenance (500 mg/m2) Q3W
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Savolitinib + Osimertinib (Experimental): 300 mg savolitinib BID plus 80 mg osimertinib QD
  Interventions: Drug: Savolitinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Savolitinib — 300 mg savolitinib (3 × 100 mg tablets twice daily) Administrative route : oral
  Other Names: AZD6094, HMPL-504, volitinib
  Arms: Savolitinib + Osimertinib
Drug: Osimertinib — 80 mg osimertinib
  (1 × 80 mg tablet once daily) Administrative route : oral
  Other Names: AZD9291, Tagrisso
  Arms: Savolitinib + Osimertinib
Drug: Pemetrexed — Pemetrexed (500 mg/m2) Administrative route : IV infusion
  Other Names: NAP
  Arms: Chemotherapy
Drug: Cisplatin — Cisplatin (75 mg/m2) or Administrative route : IV infusion
  Other Names: NAP
  Arms: Chemotherapy
Drug: Carboplatin — Carboplatin (AUC5) Administrative route : IV infusion
  Other Names: NAP
  Arms: Chemotherapy

SUMMARY:
Clinical study to investigate the efficacy and safety of savolitinib in combination with osimertinib versus platinum-based doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified, locally advanced or metastatic NSCLC who have progressed on treatment with Osimertinib.

DETAILED DESCRIPTION:
This is a multicentre, Phase III, randomised, open-label study to investigate the efficacy and safety of savolitinib administered orally in combination with osimertinib versus platinum-based doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified, locally advanced or metastatic NSCLC who have progressed on first- or second-line treatment with osimertinib as the most recent therapy.

Approximately 324 participants with EGFR mutated, MET-overexpressed and/or amplified, locally advanced or metastatic NSCLC will be randomly assigned to study intervention with 1:1 ratio.

Patients will be treated until either objective progression of disease (PD) by Response Evaluation Criteria in Solid Tumours 1.1 (RECIST 1.1) is assessed by the investigator, unacceptable toxicity occurs, consent is withdrawn, or another discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written ICF prior to any mandatory and non-mandatory study-specific procedures, sampling and analyses.
* Participant must be ≥18 years (≥ 19 years of age in South Korea) at the time of signing the informed consent. All genders are permitted.
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC which is not amenable to curative therapy.
* Must have at least one documented sensitising EGFR mutation: exon19 deletion, L858R mutation, and/or T790M.
* Documented radiologic progression on first- or second-line treatment with osimertinib as the most recent anti-cancer therapy.
* Mandatory provision of FFPE tumour tissue.
* MET overexpression and/or amplification in tumour specimen collected following progression on prior osimertinib treatment.
* Measurable disease as defined by RECIST 1.1.
* Adequate haematological, liver, renal and cardiac functions, and coagulation parameters.
* ECOG performance status of 0 or 1.

Exclusion Criteria:

* Predominant squamous NSCLC, and small cell lung cancer.
* Prior or current treatment with a third-generation EGFR-TKI other than Osimertinib.
* Prior or current treatment with savolitinib or another MET inhibitors.
* Spinal cord compression or brain metastases, unless asymptomatic and are stable.
* History or active leptomeningeal carcinomatosis.
* Unresolved toxicities from any prior therapy greater than CTCAE Grade 1 and prior platinum-therapy related Grade 2 neuropathies with the exception of alopecia and haemoglobin ≥ 9.0 g/dL.
* Active/unstable cardiac diseases currently or within the last 6 months, clinically significant ECG abnormalities, and/or factors/medications that may affect QTc intervals.
* History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement.
* Known serious active infection including, but not limited to, tuberculosis, or HIV, HBV or HCV or gastrointestinal disease.
* Receipt of live attenuated vaccine (including against COVID-19) within 30 days prior to the first dose of study intervention.
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis, which required steroid treatment, or any evidence of clinically active ILD.
* Participants currently receiving medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP)3A4 or strong inhibitors of CYP1A2.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-06-26 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) / savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified, locally advanced or metastatic NSCLC who have progressed on osimertinib. | Approximately 55 months post first subject randomized
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) /savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized.
  Defined as time from randomisation until the date of death due to any cause.
Progression-free survival (PFS) / savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed, locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
Overall Survival (OS) / savolitinib in combination with osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed by IHC, locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized
  Defined as time from randomisation until the date of death due to any cause.
Objective response rate (ORR) savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized
  ORR defined as the proportion of participants who have BOR of a CR or PR, as determined by BICR per RECIST 1.1.
Participant-reported pulmonary core symptoms / savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified, locally advanced or metastatic NSCLC who have progressed on osimertinib. | Approximately 55 months post first subject randomized
  TTD in pulmonary core symptoms (dyspnoea, cough, and chest pain) as measured by the NSCLC-SAQ.
  TTD is defined as the time from randomisation until the date of deterioration.
Pharmacokinetics (PK) of savolitinib. | 6 weeks after last patient dosed
  Plasma concentrations of savolitinib and its metabolites.
Disease control rate (DCR) / savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized
  DCR defined as the proportion of participants who have BOR of a CR, PR, or stable disease, as determined by BICR per RECIST 1.1.
Time to discontinuation of treatment (TDT) or death / savolitinib + osimertinib vs platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified locally advanced or metastatic NSCLC who have progressed on osimertinib | Approximately 55 months post first subject randomized
  TDT or death is defined as the time from date of randomisation to the earlier of the date of study intervention discontinuation or death.
Tumor shrinkage / savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized
  Tumour shrinkage defined as percentage change in tumour size in accordance with RECIST 1.1.
Duration of response (DoR) / savolitinib + osimertinib versus platinum doublet chemotherapy in participants with EGFR mutated, MET-overexpressed and/or amplified locally advanced or metastatic NSCLC who have progressed on treatment with osimertinib. | Approximately 55 months post first subject randomized
  DoR defined as the time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by BICR, or death in the absence of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Prof,MD,PhD,, Principal Investigator — Shanghai Chest Hospital, Shanghai JiaoTong University, #241 Huai Hai Road (west), Shanghai, China.
Locations (241):
- United States (12):
  - Research Site, La Jolla, California
  - Research Site, Orange City, Florida
  - Research Site, Orlando, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Evergreen Park, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Florham Park, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Canton, Ohio
  - Research Site, Nashville, Tennessee
- Argentina (9):
  - Research Site, Berazategui
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, La Rioja
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Viedma
- Australia (7):
  - Research Site, Clayton
  - Research Site, Fremantle
  - Research Site, Geelong
  - Research Site, Liverpool
  - Research Site, Southport
  - Research Site, Waratah NSW
  - Research Site, Westmead
- Austria (3):
  - Research Site, Graz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (7):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Mons
  - Research Site, Roeselare
  - Research Site, Sint-Niklaas
- Brazil (11):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Cachoeiro de Itapemirim
  - Research Site, Curitiba
  - Research Site, Ijuí
  - Research Site, Ipatinga
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Vitória
- Bulgaria (6):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- China (24):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Hankou,Wuhan
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiangfan
  - Research Site, Yichang
  - Research Site, Zhengzhou
- France (16):
  - Research Site, Angers
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Saint-Quentin
  - Research Site, Strasbourg
  - Research Site, Suresnes
- Germany (11):
  - Research Site, Berlin
  - Research Site, Chemnitz
  - Research Site, Frankfurt A. Main
  - Research Site, Gauting
  - Research Site, Homburg
  - Research Site, Immenhausen
  - Research Site, Löwenstein
  - Research Site, München
  - Research Site, Münster
  - Research Site, Stuttgart
  - Research Site, Wangen
- Greece (6):
  - Research Site, Athens
  - Research Site, Chaïdári
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Rio
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Kowloon
- Israel (6):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Be’er Ya‘aqov
  - Research Site, Hadera
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- Italy (15):
  - Research Site, Avellino
  - Research Site, Aviano
  - Research Site, Catania
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Monserrato
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Peschiera del Garda
  - Research Site, Roma
  - Research Site, Treviso
- Japan (23):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Nagasaki
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Utsunomiya
  - Research Site, Wakayama
  - Research Site, Yokohama
- Malaysia (5):
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Petaling Jaya
  - Research Site, Pulau Pinang
  - Research Site, Sabak Bernam
- Research Site, Amsterdam, Netherlands
- Philippines (8):
  - Research Site, Bacolod
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Manila
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
- Russia (4):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
- Research Site, Singapore, Singapore
- South Korea (7):
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan
- Spain (14):
  - Research Site, A Coruña
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Pontevedra
  - Research Site, Sabadell
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Switzerland (5):
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Winterthur
  - Research Site, Zurich
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Liuying
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Chanthaburi
  - Research Site, Chiang Mai
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Muang
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (8):
  - Research Site, Bristol
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newport
  - Research Site, Reading
  - Research Site, Wolverhampton
- Vietnam (3):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/335213